CLINICAL TRIAL: NCT05462600
Title: Distribution of Ventilation, Respiratory Drive and Gas Exchange: Measurements and Monitoring
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alex Pearce, Principal Investigator, University of California, San Diego
Other Study IDs: 801980
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease; Respiratory System Abnormalities; OSA; Respiratory Failure
MeSH Terms: conditions — Lung Diseases; Respiratory System Abnormalities; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BMI>24.9 kg/m2
  Interventions: Other: Position change
- BMI 18-24.9 kg/m2
  Interventions: Other: Position change

INTERVENTIONS:
Other: Position change — Distribution of ventilation, respiratory drive, pulmonary mechanics and gas exchange will be measured in 3 unique positions: prone, head of bed (HOB) flat (i.e. 0 degrees) and HOB elevated (i.e. 30 degrees).

SUMMARY:
Respiratory physiology involves a complex interplay of elements including control of breathing, respiratory drive, pulmonary mechanics, distribution of ventilation and gas exchange. Body position may also play an important role in respiratory mechanics. While effective methods exist for measuring these variables, they are typically measured in isolation rather than in combination. In pulmonary disease, decreasing mechanical stress and strain and optimizing transpulmonary pressure or the distending pressure across the lung, minimizing overdistention and collapse are central to clinical management. Obesity has a significant impact on pulmonary mechanics and is a risk factor for obstructive sleep apnea (OSA). However, our understanding of these elements is limited even in the general population. The investigators plan to use various validated methods to assess control of breathing, respiratory drive, distribution of ventilation and gas exchange to obtain a better understanding of underlying physiologic signatures in patients with and without obesity and the role of posture/position, with a secondary analysis comparing participants with and without obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Non-smokers

Exclusion Criteria:

* <18 years old
* Significant history of pulmonary disease
* Chest wall, anatomical, physical abnormalities, skin integrity issues precluding placement of electrode belt in direct contact with skin
* Skin integrity issues precluding placement of nose clips, or transcutaneous carbon dioxide monitoring
* Inability to form a seal around a mouthpiece
* Known esophageal strictures, webs, or varices (if esophageal manometry to be included)
* Known platelet count < 100,000 (if esophageal manometry to be included)
* On therapeutic anticoagulation (if esophageal manometry to be included)
* Known multidrug resistant (MDR) pulmonary infection
* Non-English language speakers
* Chronic hypoxemic respiratory failure
* Confirmed or suspected intracranial bleed, stroke, edema
* Active implants (i.e. implantable electronic devices such as pacemakers, cardioverter defibrillators or neurostimulators) or if device compatibility is in doubt
* Pregnant or lactating patients as safety and efficacy for use of EIT in such cases has not been verified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll 20 subjects with BMI 18.5-24.9 and 20 subjects with BMI 25 or more. The detailed inclusion criteria for subjects are listed below.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Distribution of ventilation | 3 hours
  Change in regional ventilation distribution (ventral/dorsal) measured through electrical impedance tomography (EIT)
Respiratory drive | 3 hours
  Respiratory drive differences will be measured by mean desaturation (change from baseline percent oxygen saturation) following breath-hold maneuvers
Respiratory drive | 3 hours
  Respiratory drive differences will be assessed by the duration of maximal breath-hold (seconds)
Respiratory drive | 3 hours
  Respiratory drive will also be assessed by measurement of occlusion pressure (cm H2O) at 100 ms (P0.1) after the initiation of an inspiratory effort against a closed circuit.

SECONDARY OUTCOMES:
Pulmonary mechanics | 3 hours
  Pulmonary mechanics will be measured by transpulmonary pressure (cmH2O)obtained from esophageal manometry (transpulmonary pressure= airway pressure- esophageal pressure)
Dead space fraction | 3 hours
  Dead space fraction will be calculated by partial pressure arterial/transcutaneous CO2 (PCO2) minus partial pressure of CO2 in mixed expired gas divided by the partial pressure of arterial/transcutaneous CO2
Ventilatory ratio | 3 hours
  Ventilatory ratio will be calculated as measured minute ventilation multiplied by the measured partial pressure of PCO2 divided (transcutaneous) by the predicted minute ventilation based on ideal body weight multiplied by the ideal PaCO2

CONTACTS AND LOCATIONS:
Overall Officials: Alex Pearce, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided